CLINICAL TRIAL: NCT04408781
Title: Clinical & Radiographic Evaluation of Split-crest Ridge Technique Versus Osseodensification Technique for Dental Implant Placement Into Narrow Alveolar Ridge
Brief Title: Management of Narrow Alveolar Ridges Via Densah-bur Versus Piezoelectric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abd el-Nabi Mohamed Amin Bilal, assistant lecturer of periodontology & oral radiology, Al-Azhar University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 104
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Knife Edge Alveolar Ridge

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ridge expansion by osseodensifcation (Experimental): Ridge expansion and osteotomy drilling by osseodensifcation in conjunction with simultaneous implant placement in narrow ridges
  Interventions: Procedure: Ridge expansion by osseodensifcation/Ridge expansion by ridge splitting
- Ridge expansion by ridge splitting (Active Comparator): Ridge expansion by ridge splitting using the piezotome in conjunction with simultaneous implant placement in narrow ridges.
  Interventions: Procedure: Ridge expansion by osseodensifcation/Ridge expansion by ridge splitting

INTERVENTIONS:
Procedure: Ridge expansion by osseodensifcation/Ridge expansion by ridge splitting — Ridge expansion by ridge splitting using the piezotome in conjunction with simultaneous implant placement in narrow ridges.
  Other Names: Ridge expansion by ridge splitting

SUMMARY:
The aim of the present study is to evaluate Clinical & radiographic evaluation of split-crest ridge technique versus osseodensification technique for dental implant placement into narrow alveolar Ridge.

DETAILED DESCRIPTION:
The aim of the study is to evaluate ridge width gain in patients with narrow alveolar ridges followingc osseodensification as compared to ridge splitting with simultaneous implant placement using CBCT.

Interventions: I. Pre-operative phase: Clinical Examination: 1. Visual examination, palpation and inspection of the entire oral and Para-oral tissues. 2. Preoperative alginate impressions for both the maxillary and the mandibular Ridges. 3. Full mouth scaling and root planing, followed by oral hygiene instructions. 4. The Bucco-Lingual/Palatal alveolar ridge width measurement at site of interest using a bone caliper. 5. Study casts will be made in order to properly evaluate the inter-arch space, occlusion type and direction of forces in regard to the site of the future implant. Radiographic Examination: 1. A panoramic radiograph for screening purposes: - estimating the residual bone height. - Verify the absence of any pathology in the bone. 2. Cone beam computed Tomography (CBCT) for Diagnostic purposes: - Detect the Bucco-lingual/palatal alveolar ridge width and height at the site of interest. - Detect approximation to any anatomical boundaries (e.g.mental foramen, maxillary sinus floor.) -Detect bone type. II. Surgical phase: All procedures will be done under strictly aseptic conditions 1. Patients will be anesthetized at the surgical site by the appropriate method using Articaine Hydrochloride 4%. 2. At the site a horizontal incision will be created, extending the entire length of the edentulous area, extending one tooth mesial and distal. Anterior and/or posterior vertical releasing incision will be made as needed. 3. Full thickness mucoperiosteal ~ap will be raised with complete exposure of the alveolar bone. 4. Bone width will be recon}rmed intrasurgically using a bone caliper. Measurements will be taken at around 1 mm below the crestal margin, to the nearest 0.5mm. Alveolar ridge width measurements will be repeated at second stage surgery. 5. A.For the intervention: 1. Drilling f bone will commence using the Pilot Drill to the desired depth (Drill speed 800-1500 rpm with copious irrigation). 2. Osseodensification drilling will begin with the narrowest Densah Bur. (Counterclockwise drill speed 800-1500 rpm with copious irrigation). If when running the bur into the osteotomy a feeling of haptic feedback of pushing up and out of the osteotomy, repetitively lifting off and reapplying pressure with a pumping motion will be applied until the desired depth is reached. 3. Densah Burs will be used sequentially in small increments. As the bur diameter increases, the bone will slowly expand to the final diameter. 4. The osteotomy final preparation diameter would be an average diameter that measures 0.5-0.8 mm smaller than the implant average diameter in soft bone, and In hard bone, diameter that measures 0.2-0.5 mm smaller than the implant average diameter. 5. Implant placement using the drill motor initially, then Finishing placement of the implant to depth with a torque-indicating wrench. 6. If < 1mm of buccal bone thickness has resulted after osseodensification, bone grafting post implant placement and complete implant coverage will be considered 5.B.For the control: 1. A bone crestal incision will be created, using the piezo-electric surgical tips. The cut will be done through the cortical bone to reach the trabecular bone. 2. One/two vertical cuts will be created by piezo-drill as needed connecting, to the crestal cut. 3. Conventional Drills will be used for osteotomy preparation by wedging it between the two plates of bone. 4. The implant with the proper length and diameter will be gradually engaged to separate the buccal and Lingual/palatal bone until full seating is achieved. 6. Cover screws will be placed on the implants. 7.Closure of the ~ap will be done by interrupted sutures using 4-0 resorbable suture materials. III. Post-operative phase: Post-operative instructions and medication: Patient is recommended to: 1. Maintain a soft diet to avoid trauma to the surgical site. 2. Place a cold compress super}cially on the skin overlying the surgical site immediately. Apply for 30 minutes, then off for 20-30 minutes. This should be done on a near continuous basis (or as much as possible) for the }first 48 hours. 3. Maintain Oral hygiene but avoid surgical site for the }rst 4 days after surgery. 4. Medications (Ferrigno et al. 2005)( Garcez-Filho et al.2015) • Augmentin* (1g tablets) will be prescribed twice daily for 5 days to avoid possibility of infection. • Ibuprofen** 600mg four times daily for one week. • Voltarene*** (75 mg injection I.M.) will be used in case of severe pain, as a rescue. • Hexitol**** 0.12% chlorhexidine mouth rinse for 2 weeks. 5. Sutures will be removed after 2 weeks 6. Final restoration will be completed after 6 months - Augmentin 1g. Medical union pharmaceuticals co. Abu Sultan, Ismailia, Egypt. **BRUFEN 600 (Ibuprofen 600 mg). Kahira Pharm. & Chem. Ind. Co., Under licence from: Abbott Laboratories. - Voltarene® 75mg/3ml (IM). Diclofenac natrium. NOVARTIS PHARMA. S.A.E. - Hexitol Chlorhexidine Hcl 125 mg / 100 ml. Arab Drug Company (ADCO).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing tooth which is needed for replacement.
2. Patients having a Bucco-lingual/palatal width of the edentulous alveolar ridge less than 6 mm. with a minimum of 3mm. residual bone width.
3. Patients having at least 11 mm residual bone height at the proposed edentulous area.
4. The recipient bed of the implant should be free from any pathological conditions.
5. No history of diagnosed bone disease or medication known to affect bone metabolism.
6. Patients who are cooperative, motivated, and has good oral hygiene.

Exclusion Criteria:

1. Patients incapable to undergoing minor oral surgical procedures.
2. Patients with insuf}cient vertical inter-arch space, upon centric occlusion, to accommodate the available restorative components.
3. Patients who have any systemic condition that may contraindicate implant therapy.
4. Patients with modifying habits affecting osteointegration for example, smoking and alcoholism.
5. Patients with parafunctional habits that can overload the implant, such as bruxism and clenching.
6. Patients with impractical expectations about the esthetic outcome of implant therapy.
7. Patients in the growth stage with mixed dentition.
8. Patients with a history of drug abuse.
9. Patients with a history of psychiatric disorder. -

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in bone width | Baseline and six month post surgically
  Cone beam computed tomography

SECONDARY OUTCOMES:
Change in Implant stability | Baseline and six month post surgically
  osstell

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed abd El-Nabi Bilal, MSC, Principal Investigator — Al-Azhar University
Locations (1):
- The Faculty of Dentistry -AL-AZHAR University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No